CLINICAL TRIAL: NCT00810667
Title: A Randomised, Double-blind, Parallel-Group, Fixed Dose Study Exploring the Efficacy and Safety of Lu AE58054 as Augmentation Therapy to Risperidone in Patients With Schizophrenia
Brief Title: Efficacy Study Exploring the Effect of Lu AE58054 as Augmentation Therapy in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12450A; 2008-001441-26 (EudraCT Number)
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Schizophrenia; Cognition
Keywords: Schizophrenia; Cognition; BACS; Risperidone; Augmentation therapy; Add-on therapy; Lu AE58054
MeSH Terms: conditions — Schizophrenia | interventions — (2-(6-fluoro-1H-indol-3-yl)-ethyl)-(3-(2,2,3,3-tetrafluoropropoxy)benzyl)amine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lu AE58054 (Experimental)
  Interventions: Drug: Lu AE58054
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lu AE58054 — twice daily oral dose (60 mg BID: total dose 120 mg/day)
  Arms: Lu AE58054
Drug: Placebo — twice daily oral dose
  Arms: Placebo

SUMMARY:
The objective of this study is to explore the efficacy, safety and cognitive properties of Lu AE58054 as augmentation therapy to risperidone in patients with schizophrenia.

DETAILED DESCRIPTION:
Lu AE58054 is a selective 5-HT6 antagonist that is currently being investigated for treatment of conditions of cognitive impairment associated with schizophrenia. Substantial experimental evidence suggests that selective 5-HT6 receptor antagonists may be effective in treating cognitive deficits since they have been shown to improve performance in various animal models of cognitive function and are known to enhance cholinergic and glutaminergic neuronal function.

Lu AE58054 has been investigated in healthy volunteers and patients with schizophrenia, is generally well tolerated and has a benign side-effect profile. Moreover, no safety concerns or issues have been identified to date.

The study is designed to provide data on the efficacy, safety and cognitive properties of Lu AE58054 as augmentation therapy to risperidone in patients with schizophrenia. Efficacy will be assessed in patients who are in a stable phase of their illness, but with a predefined minimum and maximum level of symptoms that will allow them to be included in the study. Patients will be randomly assigned to receive either the investigational medicinal product (IMP) or placebo as add-on therapy to their existing risperidone treatment.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of schizophrenia
* Man or woman, aged between 18-65
* Patient is on an optimised dose of risperidone (within 4-8 mg/day) for the treatment of schizophrenia for a minimum of 4 weeks prior to screening
* The patient has a PANSS total score between 70 and 100 (extremes included) at screening

Exclusion Criteria:

* Primary psychiatric diagnosis other than schizophrenia
* Acute exacerbation requiring hospitalisation within the last 3 months
* Clinically significant extrapyramidal symptoms
* Clinically significant cardiovascular disease, congestive heart failure, cardiac hypertrophy, arrhythmia or bradycardia
* Significant ECG abnormalities
* In concurrent treatment with drugs inhibiting the P450 enzymes system CYP2D6 and other CYP Isozymes
* Failed to respond to adequate courses of treatment with risperidone
* Treated with an antipsychotic other than risperidone within 4 weeks prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2008-11; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Efficacy effect of treatment based on the PANSS total score | 12 weeks

SECONDARY OUTCOMES:
PANSS subscales scores, CGI-S and CGI-I scores, CDSS scores, S-QoL scores, BACS, Abnormal movement scales (AIMS, BARS, SAS), ECGs, serum prolactin, pharmacokinetic assessments | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (25):
- Belgium (2):
  - BE001, Liège
  - BE005, Liège
- France (4):
  - FR002, Bordeaux
  - FR003, Brumath
  - FR001, Nîmes
  - FR006, Toulouse
- DE002, Dresden, Germany
- HK001, Hong Kong, Hong Kong
- Italy (2):
  - IT003, Brescia
  - IT004, Napoli
- Poland (11):
  - PL009, Bełchatów
  - PL006, Bialystok
  - PL002, Leszno
  - PL012, Lodz
  - PL003, Lublin
  - PL001, Lublin
  - PL010, Piekary Śląskie
  - PL004, Skorzewo
  - PL008, Torun
  - PL011, Warsaw
  - PL007, Września
- Taiwan (3):
  - TW001, Hualien City
  - TW003, Keelung
  - TW004, Tainan
- TH002, Chiang Mai, Thailand

REFERENCES:
- Available data/document: EMA EudraCT Results: 2008-001441-26 — https://www.clinicaltrialsregister.eu/ctr-search/trial/2008-001441-26/results